CLINICAL TRIAL: NCT03996707
Title: Immediate Weight-bearing Verses Non-Weight-bearing After Foot & Ankle Surgery: A Prospective Analysis
Brief Title: Immediate Weight-bearing Verses Non-Weight-bearing After Foot & Ankle Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All consented subjects were lost to follow up. P.I. stopped due to lack of interest.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Ryan McMillen, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-124JH
Record Dates: First submitted 2019-05-22; First posted 2019-06-25 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Foot and Ankle Surgery
Keywords: Ankle surgery; Foot surgery
MeSH Terms: interventions — Weight-Bearing

STUDY DESIGN:
Intervention Model Description: The investigators will be assessing the difference in two groups; immediate protected weight-bearing in a CAM walking boot vs. strict non-weight-bearing for 6 weeks following foot and ankle surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate protected weight-bearing (Other): Immediate protected weight-bearing
  Interventions: Other: Weight Bearing
- Traditional non weight bearing (Other): Strict non-weight-bearing
  Interventions: Other: Strict non-weight bearing

INTERVENTIONS:
Other: Weight Bearing — Immediate protected weight bearing in a CAM walking boot following foot & ankle surgery
  Other Names: Early Weight Bearing
  Arms: Immediate protected weight-bearing
Other: Strict non-weight bearing — Strict non weight bearing for 6 weeks following foot & ankle surgery
  Other Names: Non-weight bearing
  Arms: Traditional non weight bearing

SUMMARY:
The primary objective of this study is to determine whether immediate weight-bearing following foot and ankle surgery provides similar or superior results to the traditional non-weight-bearing post-operative course, while reducing the disuse atrophy and length of rehabilitation necessary to recover during the transition to weight-bearing following an extended course of non-weight-bearing. This will be done by way of clinical follow-up, serial radiographs and/or other appropriate imaging modalities, and patient reported outcomes by way of AOFAS and SF-36 surveys.

DETAILED DESCRIPTION:
The study is a randomized 1:1, controlled trial, prospective in nature, where participants undergoing foot and ankle surgery will be randomly placed into one of two groups; an immediate weight-bearing group or a non-weight-bearing group. The patients will be randomly placed into the study group and control group if they meet all eligibility criteria.

This study will be conducted at 5 investigative clinic sites; West Penn Hospital, Forbes Regional Hospital, Jefferson Regional Hospital, Bethel Park Surgery Center, and Monroeville Surgery. Recruitment will stop when a minimum of 230 subjects are consented.

The study duration will require 7 visits to the clinic plus a surgery day therefore will require a pre-surgical visit/screening, surgery procedural day and six outpatient post-operative visits to the clinics. The entire follow up period will occur over 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 to 89 years
2. Undergoing foot and ankle surgery
3. Must be able to read and understand English and consent for themselves

Exclusion Criteria:

1. Diagnosed peripheral neuropathy
2. Diagnosed peripheral vascular disease
3. Documented infection to the surgical extremity
4. Previous surgery to the surgical limb
5. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease which would predispose patients to poor healing and/or non-union
6. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability/Quality of Life/Satisfaction:Both Patient & Physician Assessment - American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale | Both Arms: Screening
  American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale as it pertains to the patient's ankle/foot. Pain, Function, Alignment Score 0-100, 100 being most healthy
Safety/Tolerability/Quality of Life/Satisfaction:Both Patient & Physician Assessment - American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale | Both Arms: Post-operative 6-8 weeks
  American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale as it pertains to the patient's ankle/foot. Pain, Function, Alignment Score 0-100, 100 being most healthy
Safety/Tolerability/Quality of Life/Satisfaction:Both Patient & Physician Assessment - American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale | Both Arms: Post-operative 3 month
  American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale as it pertains to the patient's ankle/foot. Pain, Function, Alignment Score 0-100, 100 being most healthy
Safety/Tolerability/Quality of Life/Satisfaction:Both Patient & Physician Assessment - American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale | Both Arms: Post-operative 12 month
  American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale as it pertains to the patient's ankle/foot. Pain, Function, Alignment Score 0-100, 100 being most healthy
Safety/Tolerability/Quality of Life/Satisfaction:Both Patient & Physician Assessment - American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale | Both Arms: Post-operative 24 month
  American Orthopaedic Foot and Ankle Score (AOFAS) Ankle-Hindfoot Scale as it pertains to the patient's ankle/foot. Pain, Function, Alignment Score 0-100, 100 being most healthy
Quality of Life/Satisfaction:Patient Report Outcome - 36 Item Short Form Survey (SF36) RAND | Both Arms: Screening
  36 Item Short Form Survey (SF36) RAND. 8 scaled scores, 0-100, 100 being most healthy
Quality of Life/Satisfaction:Patient Report Outcome - 36 Item Short Form Survey (SF36) RAND | Both Arms: Post-operative 6-8 weeks
  36 Item Short Form Survey (SF36) RAND. 8 scaled scores, 0-100, 100 being most healthy
Quality of Life/Satisfaction:Patient Report Outcome - 36 Item Short Form Survey (SF36) RAND | Both Arms: Post-operative 3 month
  36 Item Short Form Survey (SF36) RAND. 8 scaled scores, 0-100, 100 being most healthy
Quality of Life/Satisfaction:Patient Report Outcome - 36 Item Short Form Survey (SF36) RAND | Both Arms: Post-operative 12 month
  36 Item Short Form Survey (SF36) RAND. 8 scaled scores, 0-100, 100 being most healthy
Quality of Life/Satisfaction:Patient Report Outcome - 36 Item Short Form Survey (SF36) RAND | Both Arms: Post-operative 24 month
  36 Item Short Form Survey (SF36) RAND. 8 scaled scores, 0-100, 100 being most healthy

SECONDARY OUTCOMES:
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Screening
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 2-3 weeks
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 6-8 weeks
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 3 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 6 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 12 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Secondary Outcome: Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 24 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing osseous healing both clinical and radiographic evaluation.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Screening
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 2-3 weeks
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 6-8 weeks
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 3 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 6 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 12 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.
Safety/Efficacy/Tolerability - Frequency of complications during the perioperative and post-operative periods | Both arms: Post-operative 24 month
  Frequency of complications during the perioperative and post-operative periods, measured by assessing healing outcomes of soft tissue procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan L. McMillen, DPM, FACFAS, Principal Investigator — Steel Valley Orthopaedic & Sports Medicine
Locations (2):
- United States (2):
  - Steel Valley Orthopaedic and Sports Medicine, Clairton, Pennsylvania
  - The Foot & Ankle Institute/Western Pennsylvania Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Principal Investigator and Co-Investigators are part of the Allegheny Health Network and will have complete access to all data for the purpose of publication at study completion. No other outside entities are involved in this research study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03996707/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03996707/ICF_001.pdf